CLINICAL TRIAL: NCT03386994
Title: Observational Analysis on the Socio-economic Impact of IPF in Spain
Brief Title: OASIS-IPF (Idiopathic Pulmonary Fibrosis) Study
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1199-0296
Record Dates: First submitted 2017-11-16; First posted 2017-12-29 (Actual); Results first posted 2020-10-05 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-10

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Idiopathic Pulmonary Fibrosis patients: all IPF patients

SUMMARY:
Descriptive prospective non-interventional multicenter study based on newly collected data of Idiopathic Pulmonary Fibrosis patients followed-up for one year in secondary care settings (Pulmonology Services)

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients ≥ 40 years of age
* Patients diagnosed with Idiopathic Pulmonary Fibrosis (IPF) according to last ATS/ERS/JRS/ALAT IPF guideline for diagnosis and management consensus
* Written informed consent prior to participation

Exclusion Criteria:

* Inability for the patient to understand or complete the written Inform Consent or patients questionnaires or to understand Spanish
* Current participation in any clinical trial
* Patients for whom further follow-up is not possible at the enrolling site

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is planned that data of approximately 200 patients from approximately 25 sites (secondary care sites - Pulmonology services where IPF is diagnosed and managed) in Spain will be collected. All Idiopathic Pulmonary Fibrosis patients who are diagnosed with IPF and attend to a routine visit during the inclusion period and fulfill inclusion/exclusion criteria and provide informed consent to participate will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2019-09-16 (Actual); Study Completion 2019-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mireia Canals, +34607550925, Study Chair — mireia.canals@boehringer-ingelheim.com
Locations (31):
- Spain (31):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Infanta Cristina, Badajoz
  - Hospital Universitario Cruces, Barakaldo (Vizcaya)
  - H. del Mar, Barcelona
  - H. U. Vall d'Hebron, Barcelona
  - H. U. de Bellvitge, Barcelona
  - H. U. Germans Trias i Pujol, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital General Universitario Santa Lucía, Cartagena (Murcia)
  - Hospital General Universitario de Castellón, Castellon
  - H. U. de Girona Doctor Josep Trueta, Girona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Can Misses, Ibiza Town
  - Hospital Universitario Lucus Augusti, Lugo
  - H. Clínico San Carlos, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda (Madrid)
  - H. Son Llatzer, Mallorca
  - H. de Manacor, Mallorca
  - Hospital Costa del Sol, Marbella (Málaga)
  - Hospital Regional Universitario de Málaga, Málaga
  - H. Mateu Orfila, Menorca
  - Hospital Montecelo, Mourente (Pontevedra)
  - CHU de Ourense, Ourense
  - H. Central de Asturias, Oviedo
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Hospital Universitario Donostia, San Sebastián
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Hospital Sierrallana y Tres Mares, Torrelavega (Cantabria)
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Hospital Miguel Servet, Zaragoza

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Non-interventional multicenter study in Spain, based on newly collected data of patients with Idiopathic Pulmonary Fibrosis (IPF) aims to estimate the economic and social Impact of IPF according to the Forced Vital Capacity (FVC) value.
Pre-assignment Details: All patients who are diagnosed with IPF and attended to a routine visit during the inclusion period and met all of the inclusion and none of the exclusion criteria and provided informed consent to participate were included in the study. IPF-Patients were reported by subgroup (predicted FVC% at baseline) for baseline characteristics and outcome measures, to make comparisons between groups. Data on caregiver burden was collected from routine clinical care using medical records and patient´s diary.
Groups:
- All Patients With IPF - Overall Population: All patients with Idiopathic Pulmonary Fibrosis (IPF).
Period: Overall Study
Arm/Group | All Patients With IPF - Overall Population
Started (At inclusion visit (T0)) | 204
Completed (At 12 month visit (T12)) | 166
Not Completed | 38
Not completed — Lung transplant | 1
Not completed — Adverse Event | 14
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 3
Not completed — Death | 16

BASELINE CHARACTERISTICS:
Population: Evaluable Population: All participants who meet the selection criteria (no protocol deviations) and with predicted FVC% classified (in baseline visit). IPF-patients were reported by subgroups (according to predicted FVC at baseline) to make comparisons between groups.
Groups:
- IPF Patients With Predicted FVC <50% at T0 - Subgroup: All patients diagnosed with Idiopathic Pulmonary Fibrosis (IPF) and predicted Forced Vital Capacity (FVC)% value below 50% at baseline visit (T0).
  Patient group (FVC<50%, FVC 50-80%, FVC>80%) was calculated based on available patient data: Men: FVC % predicted (%)= 100 FVC/(0.678 T -0.0147 E -6.0548) Women: FVC % predicted (%)= 100 FVC /(0.0454 T -0.0211 E -2.8253) (FVC is FVC in liters, T is height in cm and E is age in years).
- IPF Patients With Predicted FVC 50-80% at T0 - Subgroup: All patients diagnosed with Idiopathic Pulmonary Fibrosis (IPF) and predicted Forced Vital Capacity (FVC)% value between 50 and 80% at baseline visit (T0).
  Patient group (FVC<50%, FVC 50-80%, FVC>80%) was calculated based on available patient data: Men: FVC % predicted (%)= 100 FVC/(0.0678 T -0.0147 E -6.0548) Women: FVC % predicted (%)= 100 FVC /(0.0454 T -0.0211 E -2.8253) (FVC is FVC in liters, T is height in cm and E is age in years).
- IPF Patients With Predicted FVC >80% at T0 - Subgroup: All patients diagnosed with Idiopathic Pulmonary Fibrosis (IPF) and predicted Forced Vital Capacity (FVC)% value above 80% at baseline visit (T0).
  Patient group (FVC<50%, FVC 50-80%, FVC>80%) was calculated based on available patient data: Men: FVC % predicted (%)= 100 FVC/(0.0678 T -0.0147 E -6.0548) Women: FVC % predicted (%)= 100 FVC /(0.0454 T -0.0211 E -2.8253) (FVC is FVC in liters, T is height in cm and E is age in years).
- Total: Total of all reporting groups
Arm/Group | IPF Patients With Predicted FVC <50% at T0 - Subgroup | IPF Patients With Predicted FVC 50-80% at T0 - Subgroup | IPF Patients With Predicted FVC >80% at T0 - Subgroup | Total
Number analyzed (Participants) | 22 | 152 | 30 | 204
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.32 (8.52) | 71.36 (7.21) | 68.33 (8.54) | 70.80 (7.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 32 | 11 | 47
  Male | 18 | 120 | 19 | 157
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Idiopathic Pulmonary Fibrosis (IPF)-Related Costs
Description: The total annual IPF-related costs were obtained as the sum of direct health costs, direct non-health costs and indirect costs. IPF-related costs were quantified for each patient over the follow-up period of 12 months. The direct health and direct non-health costs were calculated as the sum of the costs of medical visits, emergency room visits, hospital admissions, outpatient tests, non-pharmacological treatments and pharmacological treatments and the sum of transport costs, paid caregivers costs, orthopedic material costs, financial aid, and structural changes cost. The indirect costs included number of IPF related days off work and time dedicated to patient care with IPF (informal caregiver). The opportunity cost method was used to calculate informal care costs. The indirect costs were estimated by applying salary costs based on the latest data published by the Spanish Instituto Nacional de Estadística from the salary structure survey, adjusted to age.
Time Frame: 12 months. (At baseline visit (T0), at 6 months visit (T6) and at 12 month visit (T12)).
Population: Evaluable Population (cost): Evaluable Population who had data on resource use due to IPF (primary/secondary care/emergency visits, transport, hospitalization, outpatient tests, (non)-pharmacological treatment, caregivers, orthopedic material, structural changes, economic aid, lost work productivity, resource use due to acute exacerbations). IPF-patients were reported by subgroup to make comparisons between groups.
Measure: Mean (Standard Deviation); unit: Euro (€)
Arm/Group | IPF Patients With Predicted FVC <50% at T0 - Subgroup | IPF Patients With Predicted FVC 50-80% at T0 - Subgroup | IPF Patients With Predicted FVC >80% at T0 - Subgroup
Number analyzed (Participants) | 15 | 152 | 25
Euro (€)
  Total annual IPF related costs | 38923.57 (29263.42) | 22613.68 (12873.07) | 20369.94 (11955.91)
  Annual direct health IPF-related costs | 37183.17 (28465.86) | 22425.64 (12788.42) | 20195.31 (12159.89)
  Annual direct non-health related costs | 1657.63 (3148.58) | 149.25 (701.58) | 174.63 (589.53)
  Annual indirect IPF-related costs | 82.77 (320.58) | 38.79 (316.50) | 0.00 (0.00)
Statistical Analysis 1: Comparison: IPF Patients With Predicted FVC <50% at T0 - Subgroup vs IPF Patients With Predicted FVC 50-80% at T0 - Subgroup vs IPF Patients With Predicted FVC >80% at T0 - Subgroup; Test type: Other; p = 0.0002, ANOVA; Total annual IPF-related costs
Statistical Analysis 2: Comparison: IPF Patients With Predicted FVC <50% at T0 - Subgroup vs IPF Patients With Predicted FVC 50-80% at T0 - Subgroup vs IPF Patients With Predicted FVC >80% at T0 - Subgroup; Test type: Other; p = 0.0007, ANOVA; Annual direct health IPF-related costs
Statistical Analysis 3: Comparison: IPF Patients With Predicted FVC <50% at T0 - Subgroup vs IPF Patients With Predicted FVC 50-80% at T0 - Subgroup vs IPF Patients With Predicted FVC >80% at T0 - Subgroup; Test type: Other; p < 0.0001, ANOVA; Annual direct non-health IPF-related costs
Statistical Analysis 4: Comparison: IPF Patients With Predicted FVC <50% at T0 - Subgroup vs IPF Patients With Predicted FVC 50-80% at T0 - Subgroup vs IPF Patients With Predicted FVC >80% at T0 - Subgroup; Test type: Other; p = 0.6839, ANOVA; Annual indirect IPF-related costs

2. Secondary Outcome: Quality of Life (QoL) of Patients With Idiopathic Pulmonary Fibrosis (IPF) Through Saint George´s Respiratory Questionaire (SGRQ)
Description: The Quality of Life of patients with IPF according to Forced Vital Capacity (FVC)% predicted value, is assessed through SGRQ. The SGRQ is a 50-item questionaire developed to quantify the impact of the disease on the health and QoL perceived by patients with respiratory diseases. It consisted of 50 items divided into 3 scales: symptoms (frequency and severity of respiratory symptoms), activity (limitations due to dyspnoea) and impact (psychological and social functioning disorders caused by the disease). The final scores ranged from 0 (best health-related quality of life) to 100 (worse health-related quality of life). The number of participants analysed displays the number of participants with available data at the timepoint of interests.
Time Frame: 12 months. (At baseline visit (T0), at 6 month visit (T6) and at 12 month visit (T12)).
Population: Evaluable Population including participants with available data for SGRQ at T0, T6 and T12. IPF-patients were reported by subgroup to make comparisons between groups.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | IPF Patients With Predicted FVC <50% at T0 - Subgroup | IPF Patients With Predicted FVC 50-80% at T0 - Subgroup | IPF Patients With Predicted FVC >80% at T0 - Subgroup
Number analyzed (Participants) | 22 | 152 | 30
Score on a scale
  T0: number analyzed (Participants) | 21 | 143 | 29
  T0 | 48.52 (17.26) | 33.70 (17.17) | 31.97 (20.37)
  T6: number analyzed (Participants) | 13 | 118 | 24
  T6 | 43.34 (20.70) | 33.84 (19.15) | 30.68 (17.98)
  T12: number analyzed (Participants) | 12 | 109 | 22
  T12 | 41.64 (21.62) | 36.93 (19.27) | 25.38 (17.38)
Statistical Analysis 1: Comparison: IPF Patients With Predicted FVC <50% at T0 - Subgroup vs IPF Patients With Predicted FVC 50-80% at T0 - Subgroup vs IPF Patients With Predicted FVC >80% at T0 - Subgroup; Test type: Other; p = 0.0020, Kruskal-Wallis; Timepoint: T0
Statistical Analysis 2: Comparison: IPF Patients With Predicted FVC <50% at T0 - Subgroup vs IPF Patients With Predicted FVC 50-80% at T0 - Subgroup vs IPF Patients With Predicted FVC >80% at T0 - Subgroup; Test type: Other; p = 0.1385, Kruskal-Wallis; Timepoint: T6
Statistical Analysis 3: Comparison: IPF Patients With Predicted FVC <50% at T0 - Subgroup vs IPF Patients With Predicted FVC 50-80% at T0 - Subgroup vs IPF Patients With Predicted FVC >80% at T0 - Subgroup; Test type: Other; p = 0.0233, Kruskal-Wallis; Timepoint: T12

3. Secondary Outcome: Quality of Life (QoL) of Patients With Idiopathic Pulmonary Fibrosis (IPF) Through EuroQoL Visual Analogue Scale (EQ-VAS)
Description: The Quality of Life of patients with IPF according to Forced Vital Capacity (FVC)% predicted value is assessed through the EQ-VAS, which is a self-rated health status using a visual analogue scale (VAS), ranging form 0-100, with 0 = worst state of health imaginable and 100 = best state of health imaginable. The EQ-VAS is part of the EuroQoL five dimensions questionaire 5L (EQ-5D-5L).
  The number of participants analysed displays the number of participants with available data at the timepoint of interests.
Time Frame: 12 months. (At baseline visit (T0), at 6 month visit (T6) and at 12 month visit (T12)).
Population: Evaluable Population including participants with available data for EQ-VAS at T0, T6 and T12. IPF-patients were reported by subgroup to make comparisons between groups.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | IPF Patients With Predicted FVC <50% at T0 - Subgroup | IPF Patients With Predicted FVC 50-80% at T0 - Subgroup | IPF Patients With Predicted FVC >80% at T0 - Subgroup
Number analyzed (Participants) | 22 | 152 | 30
Score on a scale
  T0 | 58.41 (16.72) | 64.82 (20.43) | 66.67 (21.39)
  T6: number analyzed (Participants) | 14 | 136 | 25
  T6 | 59.29 (21.11) | 65.16 (19.02) | 68.76 (19.85)
  T12: number analyzed (Participants) | 14 | 129 | 22
  T12 | 63.93 (23.95) | 62.91 (20.34) | 71.36 (17.74)
Statistical Analysis 1: Comparison: IPF Patients With Predicted FVC <50% at T0 - Subgroup vs IPF Patients With Predicted FVC 50-80% at T0 - Subgroup vs IPF Patients With Predicted FVC >80% at T0 - Subgroup; Test type: Other; p = 0.1560, Kruskal-Wallis — Timepoint: T0
Statistical Analysis 2: Comparison: IPF Patients With Predicted FVC <50% at T0 - Subgroup vs IPF Patients With Predicted FVC 50-80% at T0 - Subgroup vs IPF Patients With Predicted FVC >80% at T0 - Subgroup; Test type: Other; p = 0.3144, Kruskal-Wallis — Timepoint: T6
Statistical Analysis 3: Comparison: IPF Patients With Predicted FVC <50% at T0 - Subgroup vs IPF Patients With Predicted FVC 50-80% at T0 - Subgroup vs IPF Patients With Predicted FVC >80% at T0 - Subgroup; Test type: Other; p = 0.2019, Kruskal-Wallis — Timepoint: T12

4. Secondary Outcome: Quality of Life (QoL) of Patients With Idiopathic Pulmonary Fibrosis (IPF), Through Barthel Index
Description: The Quality of Life of patients with IPF according to Forced Vital Capacity (FVC)% predicted value is assessed through the Barthel Index.
  Barthel Index were used to score the ability of a participant to care for himself. It consists of 10 items, the values assigned to each item are based on time and amount of actual physical assistance required if a participant is unable to perform the activity. The final score ranges from 0 and 100. Participant scoring 100 is continent, feeds himself, dresses himself, gets up out of bed and chairs, bathes himself, walks at least a block, and can ascend and descend stairs.
  The number of participants analysed displays the number of participants with available data at the timepoint of interests.
Time Frame: 12 months. (At baseline visit (T0), at 6 month visit (T6) and at 12 month visit (T12)).
Population: Evaluable Population including participants with available data for Barthel Index at T0, T6 and T12. IPF-patients were reported by subgroup to make comparisons between groups.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | IPF Patients With Predicted FVC <50% at T0 - Subgroup | IPF Patients With Predicted FVC 50-80% at T0 - Subgroup | IPF Patients With Predicted FVC >80% at T0 - Subgroup
Number analyzed (Participants) | 22 | 152 | 30
Score on a scale
  T0 | 92.95 (10.76) | 97.50 (7.68) | 97.67 (5.68)
  T6: number analyzed (Participants) | 12 | 138 | 26
  T6 | 91.25 (12.08) | 95.94 (11.21) | 96.35 (8.19)
  T12: number analyzed (Participants) | 14 | 129 | 22
  T12 | 91.79 (15.76) | 95.74 (12.66) | 96.59 (12.85)
Statistical Analysis 1: Comparison: IPF Patients With Predicted FVC <50% at T0 - Subgroup vs IPF Patients With Predicted FVC 50-80% at T0 - Subgroup vs IPF Patients With Predicted FVC >80% at T0 - Subgroup; Test type: Other; p = 0.0075, Kruskal-Wallis — Timepoint: T0
Statistical Analysis 2: Comparison: IPF Patients With Predicted FVC <50% at T0 - Subgroup vs IPF Patients With Predicted FVC 50-80% at T0 - Subgroup vs IPF Patients With Predicted FVC >80% at T0 - Subgroup; Test type: Other; p = 0.0361, Kruskal-Wallis — Timepoint: T6
Statistical Analysis 3: Comparison: IPF Patients With Predicted FVC <50% at T0 - Subgroup vs IPF Patients With Predicted FVC 50-80% at T0 - Subgroup vs IPF Patients With Predicted FVC >80% at T0 - Subgroup; Test type: Other; p = 0.4794, Kruskal-Wallis — Timepoint: T12

5. Secondary Outcome: Number of Idiopathic Pulmonary Fibrosis (IPF)-Patients With Acute Exacerbations Along One Year
Description: Number of IPF-patients with acute exacerbations according to Forced Vital Capacity (FVC)% that occured along one year.
  Acute exacerbation is defined as an acute, clinically significant respiratory deterioration characterized by evidence of new widespread alveolar abnormality.
Time Frame: 12 months. (At baseline visit (T0), at 6 month visit (T6) and at 12 month visit (T12)).
Population: Evaluable Population: All patients who met the selection criteria (no protocol deviations) and with predicted FVC% classified. IPF-patients were reported by subgroup to make comparisons between groups.
Measure: Number; unit: Participants
Arm/Group | IPF Patients With Predicted FVC <50% at T0 - Subgroup | IPF Patients With Predicted FVC 50-80% at T0 - Subgroup | IPF Patients With Predicted FVC >80% at T0 - Subgroup
Number analyzed (Participants) | 22 | 152 | 30
Participants | 6 | 13 | 3
Statistical Analysis 1: Comparison: IPF Patients With Predicted FVC <50% at T0 - Subgroup vs IPF Patients With Predicted FVC 50-80% at T0 - Subgroup vs IPF Patients With Predicted FVC >80% at T0 - Subgroup; Test type: Other; p = 0.0333, Fisher Exact

6. Secondary Outcome: Total Annual Acute Exacerbation-related Costs
Description: The total annual acute exacerbation-related costs were obtained as the sum of direct and indirect costs for each patient over the follow-up period of 12 months.
  For estimation of costs the following variables were used: Acute exacerbation related resource use for direct cost estimation: primary and secondary care visits, emergency visits (primary care and hospital), hospitalizations, ICU with and without intubation (qualitative analysis), outpatient tests and other examinations, use of transport, use of formal caregiver, pharmacological and non-pharmacological treatments (except treatments administered in hospitalization), orthopedic material, formal social services, economic aid and structural adaptations. Acute exacerbation related resource use for indirect cost estimation: patients' days off work and informal caregiver.
Time Frame: 12 months. (At baseline visit (T0), at 6 months visit (T6) at 12 month visit (T12)).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Euro (€)
Arm/Group | IPF Patients With Predicted FVC <50% at T0 - Subgroup | IPF Patients With Predicted FVC 50-80% at T0 - Subgroup | IPF Patients With Predicted FVC >80% at T0 - Subgroup
Number analyzed (Participants) | 15 | 140 | 25
Euro (€) | 600.40 (1586.20) | 819.28 (3827.04) | 142.17 (703.24)

7. Secondary Outcome: Idiopathic Pulmonary Fibrosis (IPF)-Related Costs by Forced Vital Capacity (FVC) Decline - Overall FVC Patient Group
Description: Economic Impact of IPF in adult patients through the estimation annual direct and indirect costs associated with the disease (€/year) from a social perspective by FVC decline according to predicted FVC%.
  FVC decline is calculated: FVC% (T12)- FVC%(T0)).
  In order to estimate the direct and indirect costs according to FVC decline the following variable were described:
  FVC predicted along the study. Men: FVC % predicted (%) = 100 FVC / (0.0678 T - 0.0147 E - 6.0548) Women: FVC % predicted (%) = 100 FVC / (0.0454 T - 0.0211 E - 2.8253)
  (FVC is FVC in liters, T is height in cm and E is age in years)
  The calculated variable was stratified into the following subgroups between T0 and T12:
  ≤-10%; from -10% to -5%; >-5%
Time Frame: 12 months. (At baseline visit (T0) and at 12 month visit (T12)).
Population: Evaluable Population (cost) including participants with FVC decline between T0 and T12 (paired data) - Overall FVC Patient Group.
Measure: Mean (Standard Deviation); unit: Euro (€)
Groups:
- <-10% FVC Decline: IPF patients with FVC decline less than -10%.
- From -10 to -5% FVC Decline: IPF patients with FVC decline from -10% to -5%.
- >-5% FVC Decline: IPF patients with FVC decline more than -5%.
Arm/Group | <-10% FVC Decline | From -10 to -5% FVC Decline | >-5% FVC Decline
Number analyzed (Participants) | 24 | 31 | 85
Euro (€)
  Total annual IPF-related costs | 22261.30 (14568.38) | 20986.06 (10864.08) | 26171.47 (17009.81)
  Annual direct health IPF-related costs | 21926.97 (14418.41) | 20939.38 (10847.61) | 25818.15 (16606.63)
  Annual direct non-health IPF-related costs | 331.35 (918.61) | 0.00 (0.00) | 349.66 (1511.20)
  Annual indirect IPF-related costs | 2.99 (14.63) | 46.68 (185.74) | 3.65 (24.86)
Statistical Analysis 1: Comparison: <-10% FVC Decline vs From -10 to -5% FVC Decline vs >-5% FVC Decline; Test type: Other; p = 0.4711, ANOVA; Total annual IPF-related costs
Statistical Analysis 2: Comparison: <-10% FVC Decline vs From -10 to -5% FVC Decline vs >-5% FVC Decline; Test type: Other; p = 0.4095, ANOVA; Annual direct health IPF-related costs
Statistical Analysis 3: Comparison: <-10% FVC Decline vs From -10 to -5% FVC Decline vs >-5% FVC Decline; Test type: Other; p = 0.0435, ANOVA; Annual direct non-health IPF-related costs
Statistical Analysis 4: Comparison: <-10% FVC Decline vs From -10 to -5% FVC Decline vs >-5% FVC Decline; Test type: Other; p = 0.5479, ANOVA; Annual indirect IPF-related costs

8. Secondary Outcome: Idiopathic Pulmonary Fibrosis (IPF)-Related Costs by Forced Vital Capacity (FVC) Decline - Subgroup: Predicted FVC<50% at T0
Description: Economic Impact of IPF in adult patients through the estimation annual direct and indirect costs associated with the disease (€/year) from a social perspective by FVC decline according to predicted FVC%.
  FVC decline is calculated: FVC% (T12)- FVC%(T0)).
  In order to estimate the direct and indirect costs according to FVC decline the following variable were described:
  FVC predicted along the study. Men: FVC % predicted (%) = 100 FVC / (0.0678 T - 0.0147 E - 6.0548) Women: FVC % predicted (%) = 100 FVC / (0.0454 T - 0.0211 E - 2.8253)
  (FVC is FVC in liters, T is height in cm and E is age in years)
  The calculated variable was stratified into the following subgroups between T0 and T12:
  ≤-10%; from -10% to -5%; >-5%
  Results are reported for participants with predicted FVC <50% at baseline.
Time Frame: 12 months. (At baseline visit (T0) and at 12 month visit (T12)).
Population: Evaluable Population (cost) including participants with FVC decline between T0 and T12 (paired data) - Subgroup with predicted FVC <50% at T0.
Measure: Mean (Standard Deviation); unit: Euro (€)
Groups:
- <-10% FVC Decline: IPF patients with less than -10% FVC decline.
- From -10% to -5% FVC Decline: IPF patients with FVC decline from -10% to - 5%.
Arm/Group | <-10% FVC Decline | From -10% to -5% FVC Decline | >-5% FVC Decline
Number analyzed (Participants) | 0 | 0 | 9
Euro (€)
  Total annual IPF-related costs |  |  | 48035.14 (32937.16)
  Annual direct health IPF-related costs |  |  | 45646.56 (32130.57)
  Annual direct non-health related costs |  |  | 2388.58 (3902.02)
  Annual indirect IPF-related costs |  |  | 0.00 (0.00)

9. Secondary Outcome: Idiopathic Pulmonary Fibrosis (IPF)-Related Costs by Forced Vital Capacity (FVC) Decline - Subgroup: Predicted FVC 50-80% at T0
Description: Economic Impact of IPF in adult patients through the estimation annual direct and indirect costs associated with the disease (€/year) from a social perspective by FVC decline according to predicted FVC%.
  FVC decline is calculated: FVC% (T12)- FVC%(T0)).
  In order to estimate the direct and indirect costs according to FVC decline the following variable were described:
  Men: FVC % predicted (%) = 100 FVC / (0.0678 T - 0.0147 E - 6.0548) Women: FVC % predicted (%) = 100 FVC / (0.0454 T - 0.0211 E - 2.8253)
  (FVC is FVC in liters, T is height in cm and E is age in years)
  The calculated variable was stratified into the following subgroups between T0 and T12:
  ≤-10%; from -10% to -5%; >-5%
  Results are reported for participants with predicted FVC 50-80% at baseline.
Time Frame: 12 months. (At baseline visit (T0) and at 12 month visit (T12)).
Population: Evaluable Population (cost) including participants with FVC decline between T0 and T12 (paired data) - Subgroup predicted FVC 50-80% at T0.
Measure: Mean (Standard Deviation); unit: Euro (€)
Groups:
- From -10% to -5% FVC Decline: IPF patients with FVC decline from -10% to -5%
Arm/Group | <-10% FVC Decline | From -10% to -5% FVC Decline | >-5% FVC Decline
Number analyzed (Participants) | 21 | 26 | 64
Euro (€)
  Total annual IPF-related costs | 24208.51 (14372.38) | 20546.19 (11062.92) | 23539.60 (11999.95)
  Annual direct health IPF-related costs | 23826.41 (14251.63) | 20490.53 (11041.18) | 23450.00 (12009.78)
  Annual direct non-healt IPF-related costs | 378.68 (975.49) | 0.00 (0.00) | 84.75 (574.20)
  Annual indirect IPF-related costs | 3.41 (15.64) | 55.66 (202.19) | 4.85 (28.60)
Statistical Analysis 1: Comparison: <-10% FVC Decline vs From -10% to -5% FVC Decline vs >-5% FVC Decline; Test type: Other; p = 0.7486, ANOVA; Total annual IPF-related costs
Statistical Analysis 2: Comparison: <-10% FVC Decline vs From -10% to -5% FVC Decline vs >-5% FVC Decline; Test type: Other; p = 0.7652, ANOVA; Annual direct health IPF-related costs
Statistical Analysis 3: Comparison: <-10% FVC Decline vs From -10% to -5% FVC Decline vs >-5% FVC Decline; Test type: Other; p = 0.0037, ANOVA; Annual direct non-health IPF-related costs
Statistical Analysis 4: Comparison: <-10% FVC Decline vs From -10% to -5% FVC Decline vs >-5% FVC Decline; Test type: Other; p = 0.6119, ANOVA; Annual indirect IPF-related costs

10. Secondary Outcome: Idiopathic Pulmonary Fibrosis (IPF)-Related Costs by Forced Vital Capacity (FVC) Decline - Subgroup: Predicted FVC>80% at T0
Description: Economic Impact of IPF in adult patients through the estimation annual direct and indirect costs associated with the disease (€/year) from a social perspective by FVC decline according to predicted FVC%.
  FVC decline is calculated: FVC% (T12)- FVC%(T0)).
  In order to estimate the direct and indirect costs according to FVC decline the following variable were described:
  Men: FVC % predicted (%) = 100 FVC / (0.0678 T - 0.0147 E - 6.0548) Women: FVC % predicted (%) = 100 FVC / (0.0454 T - 0.0211 E - 2.8253)
  (FVC is FVC in liters, T is height in cm and E is age in years)
  The calculated variable was stratified into the following subgroups between T0 and T12:
  ≤-10%; from -10% to -5%; >-5%
  Results are reported for participants with predicted FVC > 80% at baseline.
Time Frame: 12 months. (At baseline visit (T0) and at 12 month visit (T12)).
Population: Evaluable Population (cost) including participants with FVC decline between T0 and T12 (paired data) - Subgroup with predicted FVC >80% at T0.
Measure: Mean (Standard Deviation); unit: Euro (€)
Arm/Group | <-10% FVC Decline | From -10% to -5% FVC Decline | >-5% FVC Decline
Number analyzed (Participants) | 3 | 5 | 12
Euro (€)
  Total annual IPF-related costs | 8630.88 (7522.53) | 23273.38 (10606.04) | 23810.32 (12580.11)
  Annual direct health IPF-related costs | 8630.88 (7522.53) | 23273.38 (10606.04) | 23576.99 (13010.66)
  Annual direct non-health IPF-related costs | 0.00 (0.00) | 0.00 (0.00) | 233.33 (808.29)
  Annual indirect IPF-related costs | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
Statistical Analysis 1: Comparison: <-10% FVC Decline vs From -10% to -5% FVC Decline vs >-5% FVC Decline; Test type: Other; p = 0.1581, ANOVA; Total annual IPF-related costs
Statistical Analysis 2: Comparison: <-10% FVC Decline vs From -10% to -5% FVC Decline vs >-5% FVC Decline; Test type: Other; p = 0.1581, ANOVA; Annual direct health IPF-related costs
Statistical Analysis 3: Comparison: <-10% FVC Decline vs From -10% to -5% FVC Decline vs >-5% FVC Decline; Test type: Other; p = 0.7165, ANOVA; Annual direct non-health IPF-related costs
Statistical Analysis 4: Comparison: <-10% FVC Decline vs From -10% to -5% FVC Decline vs >-5% FVC Decline; Test type: Other; p = 1.0000, ANOVA; Annual indirect IPF-related costs

11. Secondary Outcome: Absolute Change in Saint George´s Respiratory Questionaire (SGRQ) Score From Baseline Visit (T0) to 12 Month Visit (T12) by Forced Vital Capacity (FVC) Decline - Overall FVC Patient Group
Description: Absolute Change in SGRQ score by FVC decline according to predicted FVC% from baseline visit (T0) to 12 month visit (T12).
  The SGRQ is a 50-item questionaire developed to quantify the impact of the disease on the health and QoL perceived by patients with respiratory diseases. It consisted of 50 items divided into 3 scales: symptoms, activity and impact. The final scores ranged from 0 (best health-related quality of life) to 100 (worse health-related quality of life).
  FVC decline: FVC% (T12)- FVC%(T0)
  In order to estimate the Quality of Life according to FVC decline the following variable were described:
  FVC % predicted along the study:. Men: FVC % predicted (%) = 100 FVC / (0.0678 T - 0.0147 E - 6.0548) Women: FVC % predicted (%) = 100 FVC / (0.0454 T - 0.0211 E - 2.8253)
  (FVC is FVC in liters, T is height in cm and E is age in years).
  The calculated variable was stratified into the following subgroups between T0 and T12:
  ≤-10%; from -10% to -5%; >-5%
Time Frame: 12 months. (At baseline visit (T0) and at 12 month visit (T12)).
Population: Evaluable Population including participants with FVC decline between T0 and T12 (paired data) and with SGRQ values at T0 and T12 - Overall FVC patient group.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | <-10% FVC Decline | From -10% to -5% FVC Decline | >-5% FVC Decline
Number analyzed (Participants) | 18 | 25 | 72
Score on a scale | 8.49 (17.16) | 3.20 (11.71) | 0.23 (13.11)
Statistical Analysis 1: Comparison: <-10% FVC Decline vs From -10% to -5% FVC Decline vs >-5% FVC Decline; Test type: Other; p = 0.0733, Kruskal-Wallis

12. Secondary Outcome: Absolute Change in Saint George´s Respiratory Questionaire (SGRQ) Score From Baseline Visit (T0) to 12 Month Visit (T12) by Forced Vital Capacity (FVC) Decline - Subgroup: Predicted FVC<50% at T0
Description: Absolute Change in SGRQ score by FVC decline according to predicted FVC% from baseline visit (T0) to 12 month visit (T12).
  The SGRQ is a 50-item questionaire developed to quantify the impact of the disease on the health and QoL perceived by patients with respiratory diseases. It consisted of 50 items divided into 3 scales: symptoms, activity and impact. The final scores ranged from 0 (best health-related quality of life) to 100 (worse health-related quality of life).
  FVC decline: FVC% (T12)- FVC%(T0)
  In order to estimate SGRQ according to FVC decline the following variable were described:
  Men: FVC % predicted (%) = 100 FVC / (0.0678 T - 0.0147 E - 6.0548) Women: FVC % predicted (%) = 100 FVC / (0.0454 T - 0.0211 E - 2.8253)
  (FVC is FVC in liters, T is height in cm and E is age in years).
  The calculated variable was stratified into the following subgroups between T0 and T12:
  ≤-10%; from -10% to -5%; >-5%
  Results are reported for participants with predicted FVC<50% at baseline.
Time Frame: 12 months. (At baseline visit (T0) and at 12 month visit (T12)).
Population: Evaluable Population including participants with FVC decline between T0 and T12 (paired data) and with SGRQ values at T0 and T12 - Subgroup with predicted FVC <50% at T0.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | <-10% FVC Decline | From -10% to -5% FVC Decline | >-5% FVC Decline
Number analyzed (Participants) | 0 | 0 | 7
Score on a scale |  |  | -14.93 (29.03)

13. Secondary Outcome: Absolute Change in Saint George´s Respiratory Questionaire (SGRQ) Score From Baseline Visit (T0) to 12 Month Visit (T12) by Forced Vital Capacity (FVC) Decline - Subgroup: Predicted FVC 50-80% at T0
Description: Absolute Change in SGRQ score by FVC decline according to predicted FVC% from baseline visit (T0) to 12 month visit (T12).
  The SGRQ is a 50-item questionaire developed to quantify the impact of the disease on the health and QoL perceived by patients with respiratory diseases. It consisted of 50 items divided into 3 scales: symptoms (frequency and severity of respiratory symptoms), activity (limitations due to dyspnoea) and impact (psychological and social functioning disorders caused by the disease). The final scores ranged from 0 (best health-related quality of life) to 100 (worse health-related quality of life).
  FVC decline: FVC% (T12)- FVC%(T0)
  Results are reported for participants with predicted FVC 50-80% at baseline.
Time Frame: 12 months (At baseline visit (T0) and at 12 month visit (T12)).
Population: Evaluable Population including participants with FVC decline between T0 and T12 (paired data) and with SGRQ values at T0 and T12 - Subgroup with predicted FVC 50-80% at T0.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | <-10% FVC Decline | From -10% to -5% FVC Decline | >-5% FVC Decline
Number analyzed (Participants) | 15 | 21 | 53
Score on a scale | 12.58 (14.02) | 2.20 (12.16) | 2.16 (9.62)
Statistical Analysis 1: Comparison: <-10% FVC Decline vs From -10% to -5% FVC Decline vs >-5% FVC Decline; Test type: Other; p = 0.0207, Kruskal-Wallis

14. Secondary Outcome: Absolute Change in Saint George´s Respiratory Questionaire (SGRQ) Score From Baseline Visit (T0) to 12 Month Visit (T12) by Forced Vital Capacity (FVC) Decline - Subgroup: Predicted FVC>80% at T0
Description: Absolute Change in SGRQ score by FVC decline according to predicted FVC% from baseline visit (T0) to 12 month visit (T12).
  The SGRQ is a 50-item questionaire developed to quantify the impact of the disease on the health and QoL perceived by patients with respiratory diseases. It consisted of 50 items divided into 3 scales: symptoms (frequency and severity of respiratory symptoms), activity (limitations due to dyspnoea) and impact (psychological and social functioning disorders caused by the disease). The final scores ranged from 0 (best health-related quality of life) to 100 (worse health-related quality of life).
  FVC decline: FVC% (T12)- FVC%(T0)
  Results are reported for participants with predicted FVC >80% at baseline.
Time Frame: 12 months. (At baseline visit (T0) and at 12 month visit (T12)).
Population: Evaluable Population including participants with FVC decline between T0 and T12 (paired data) and with SGRQ values at T0 and T12 - Subgroup with predicted FVC >80% at T0.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | <-10% FVC Decline | From -10% to -5% FVC Decline | >-5% FVC Decline
Number analyzed (Participants) | 3 | 4 | 12
Score on a scale | -11.97 (19.38) | 8.43 (8.32) | 0.56 (6.93)
Statistical Analysis 1: Comparison: <-10% FVC Decline vs From -10% to -5% FVC Decline vs >-5% FVC Decline; Test type: Other; p = 0.0942, Kruskal-Wallis

15. Secondary Outcome: Absolute Change in EuroQoL Visual Analogue Scale (EQ-VAS) From Baseline Visit (T0) to 12 Month Visit (T12) by Forced Vital Capacity (FVC) Decline- Overall FVC Patient Group
Description: Absolute Change in EQ-VAS score by FVC decline according to predicted FVC% from baseline visit (T0) to 12 month visit (T12). The EQVAS is a self-rated health status using a VAS (0-100), with 0= worst state of health imaginable and 100= best state of health imaginable. The EQ-VAS records the subject's perceptions of their own current overall health.
  FVC decline: FVC% (T12)- FVC%(T0)
  In order to estimate the EQ-VAS according to FVC decline the following variable were described:
  FVC % predicted along the study:
  Men: FVC % predicted (%) = 100 FVC / (0.0678 T - 0.0147 E - 6.0548) Women: FVC % predicted (%) = 100 FVC / (0.0454 T - 0.0211 E - 2.8253)
  (FVC is FVC in liters, T is height in cm and E is age in years)
  The calculated variable was stratified into the following subgroups between T0 and T12:
  ≤-10%; from -10% to -5%; >-5%
Time Frame: 12 months. (At baseline visit (T0) and at 12 month visit (T12)).
Population: Evaluable Population including participants with FVC decline between T0 and T12 (paired data) and with EQ-VAS values at T0 and T12 - Overall FVC Patient Group.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | <-10% FVC Decline | From -10% to -5% FVC Decline | >-5% FVC Decline
Number analyzed (Participants) | 24 | 31 | 85
Score on scale | -8.96 (17.74) | -6.16 (18.69) | -0.04 (14.79)
Statistical Analysis 1: Comparison: <-10% FVC Decline vs From -10% to -5% FVC Decline vs >-5% FVC Decline; Test type: Other; p = 0.0747, Kruskal-Wallis

16. Secondary Outcome: Absolute Change in EuroQoL Visual Analogue Scale (EQ-VAS) From Baseline Visit (T0) to 12 Month Visit (T12) by Forced Vital Capacity (FVC) Decline - Subgroup: Predicted FVC<50% at T0
Description: Absolute Change in EQ-VAS score by FVC decline according to predicted FVC% from baseline visit (T0) to 12 month visit (T12).
  The EQVAS is a self-rated health status using a VAS (0-100), with 0= worst state of health imaginable and 100= best state of health imaginable. The EQ-VAS records the subject's perceptions of their own current overall health.
  FVC decline: FVC% (T12)- FVC%(T0)
  In order to estimate the EQ-VAS according to FVC decline the following variable were described:
  FVC % predicted along the study:
  Men: FVC % predicted (%) = 100 FVC / (0.0678 T - 0.0147 E - 6.0548) Women: FVC % predicted (%) = 100 FVC / (0.0454 T - 0.0211 E - 2.8253) (FVC is FVC in liters, T is height in cm and E is age in years)
  The calculated variable was stratified into the following subgroups between T0 and T12:
  ≤-10%; from -10% to -5%; >-5% Results are reported for participants with predicted FVC<50% at baseline.
Time Frame: 12 months. (At baseline visit (T0) and at 12 month visit (T12)).
Population: Evaluable Population including participants with FVC decline between T0 and T12 (paired data) and with EQ-VAS values at T0 and T12 - Subgroup with predicted FVC <50% at T0.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | <-10% FVC Decline | From -10% to -5% FVC Decline | >-5% FVC Decline
Number analyzed (Participants) | 0 | 0 | 9
Score on scale |  |  | 13.89 (13.41)

17. Secondary Outcome: Absolute Change in EuroQoL Visual Analogue Scale (EQ-VAS) From Baseline Visit (T0) to 12 Month Visit (T12) by Forced Vital Capacity (FVC) Decline- Subgroup: Predicted FVC 50-80% at T0
Description: Absolute Change in EQ-VAS score by FVC decline according to predicted FVC% from baseline visit (T0) to 12 month visit (T12).
  The EQVAS is a self-rated health status using a VAS (0-100), with 0= worst state of health imaginable and 100= best state of health imaginable. The EQ-VAS records the subject's perceptions of their own current overall health.
  FVC decline: FVC% (T12)- FVC%(T0)
  In order to estimate the EQ-VAS according to FVC decline the following variable were described:
  FVC % predicted along the study:. Men: FVC % predicted (%) = 100 FVC / (0.0678 T - 0.0147 E - 6.0548) Women: FVC % predicted (%) = 100 FVC / (0.0454 T - 0.0211 E - 2.8253) (FVC is FVC in liters, T is height in cm and E is age in years)
  The calculated variable was stratified into the following subgroups between T0 and T12:
  ≤-10%; from -10% to -5%; >-5% Results are reported for participants with predicted FVC 50-80% at baseline.
Time Frame: 12 months. (At baseline visit (T0) and at 12 month visit (T12)).
Population: Evaluable Population including participants with FVC decline between T0 and T12 (paired data) and with EQ-VAS values at T0 and T12 - Subgroup with predicted FVC 50-80% at T0.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | <-10% FVC Decline | From -10% to -5% FVC Decline | >-5% FVC Decline
Number analyzed (Participants) | 21 | 26 | 64
Score on scale | -10.48 (18.21) | -6.96 (20.15) | -1.45 (14.77)
Statistical Analysis 1: Comparison: <-10% FVC Decline vs From -10% to -5% FVC Decline vs >-5% FVC Decline; Test type: Other; p = 0.1282, Kruskal-Wallis

18. Secondary Outcome: Absolute Change in EuroQoL Visual Analogue Scale (EQ-VAS) From Baseline Visit (T0) to 12 Month Visit (T12) by Forced Vital Capacity (FVC) Decline - Subgroup: Predicted FVC>80% at T0
Description: Absolute Change in EQ-VAS score by FVC decline according to predicted FVC% from baseline visit (T0) to 12 month visit (T12).
  The EQVAS is a self-rated health status using a VAS (0-100), with 0= worst state of health imaginable and 100= best state of health imaginable. The EQ-VAS records the subject's perceptions of their own current overall health.
  FVC decline: FVC% (T12)- FVC%(T0)
  In order to estimate the EQ-VAS according to FVC decline the following variable were described:
  FVC % predicted along the study:. Men: FVC % predicted (%) = 100 FVC / (0.0678 T - 0.0147 E - 6.0548) Women: FVC % predicted (%) = 100 FVC / (0.0454 T - 0.0211 E - 2.8253) (FVC is FVC in liters, T is height in cm and E is age in years)
  The calculated variable was stratified into the following subgroups between T0 and T12:
  ≤-10%; from -10% to -5%; >-5% Results are reported for participants with predicted FVC>80% at baseline.
Time Frame: 12 months. (At baseline visit (T0) and at 12 month visit (T12)).
Population: Evaluable Population including participants with FVC decline between T0 and T12 (paired data) and with EQ-VAS values at T0 and T12 - Subgroup with predicted FVC >80% at T0.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | <-10% FVC Decline | From -10% to -5% FVC Decline | >-5% FVC Decline
Number analyzed (Participants) | 3 | 5 | 12
Score on scale | 1.67 (10.41) | -2.00 (7.58) | -2.92 (10.54)
Statistical Analysis 1: Comparison: <-10% FVC Decline vs From -10% to -5% FVC Decline vs >-5% FVC Decline; Test type: Other; p = 0.7471, Kruskal-Wallis

19. Secondary Outcome: Impact of Disease on the Patients Caregiver Through Zarit Burden Interview Questionaire
Description: Caregivers of IPF patients were asked to complete the Zarit Burden Interview. It is a self-report measure. The revised version contains 22 items. Each item on the interview is a statement which the caregiver is asked to endorse using a 5-point scale. Response options, in the Spanish version, range from 0 (never) to 4 (nearly always).
  The final score ranges from 0 to 88. A higher score implies a greater burden (≤ 21: Little or no burden; 22-40: mild to moderate burden; 41-60: moderate to severe burden; ≥ 61: severe burden).
Time Frame: 12 months. (At baseline visit (T0), at 6 month visit (T6), at 12 month visit (T12)).
Population: Caregivers who have signed the specific written informed consent.
Measure: Mean (Standard Deviation); unit: Score an a scale
Groups:
- Caregivers: Caregivers of patients with Idiopathic Pulmonary Fibrosis.
Arm/Group | Caregivers
Number analyzed (Participants) | 37
Score an a scale
  T0 | 23.59 (15.81)
  T6: number analyzed (Participants) | 26
  T6 | 22.50 (17.99)
  T12: number analyzed (Participants) | 25
  T12 | 22.08 (19.45)

ADVERSE EVENTS:
Time Frame: From signing informed consent until end of study, up to 12 months.
Description: For all-cause mortality and serious adverse events the safety population (All screened patients with informed consent prior to participation) was used. Other Adverse events were reported only for patients with at least one dose of OFEV® (OFEV® Population), as defined in the study report. Please note that the number of deaths reported in all-cause mortality is higher than reported in the participant flow due to a number of participants dying after discontinuing the study.
Arm/Group | All Patients With IPF - Overall Population
All-Cause Mortality (participants affected / at risk) | 30/204
Serious Adverse Events (participants affected / at risk) | 31/204
Other Adverse Events (participants affected / at risk) | 12/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients With IPF - Overall Population (N=204)
Acute myocardial infarction (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Death (General disorders) | 3
Disease progression (General disorders) | 3
Bronchitis (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Completed suicide (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 6
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Solid organ transplant (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients With IPF - Overall Population (N=89)
Diarrhoea (Gastrointestinal disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-10-30): https://cdn.clinicaltrials.gov/large-docs/94/NCT03386994/SAP_001.pdf
  • Study Protocol (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/94/NCT03386994/Prot_002.pdf